CLINICAL TRIAL: NCT00842647
Title: Diagnosis of Hepatic Tumors in Cirrhosis: Prospective Validation of the Noninvasive Diagnostic Criteria for Hepatocellular Carcinoma
Acronym: HCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Ministry of Health, China (Other Government)
Responsible Party: Cancer Center, Sun Yat-sen University, Cancer Center, Sun Yat-sen University
Other Study IDs: HCC05
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Sensitivity; specificity; positive rate; negative rate
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study prospectively evaluates the accuracy of the noninvasive diagnostic criteria for hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. All the patients who receive hepatomy in our department
2. Diagnose as HCC
3. Diagnosis of HCC is confirmed by noninvasive criteria for HCC as used by the American Association for the Study of the Liver guidelines
4. No history of previous treatments
5. No pathological diagnosis before treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between July 2006 and July 2009
  1. All the patients who receive hepatomy in our department
  2. Diagnose as HCC
  3. Diagnosis of HCC is confirmed by noninvasive criteria for HCC as used by the American Association for the Study of the Liver guidelines
  4. No history of previous treatments
  5. No pathological diagnosis before treatment
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2006-07; Primary Completion 2009-07 (Estimated); Study Completion 2009-08 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hepatobilliary Surgery, Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Bruix J, Sherman M. Practice Guidelines Committee, American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma. Hepatology. 2005;42:1208-1236 Parkin DM, Bray F, Ferlay J, Pisani P. Global cancer statistics, 2002. CA Cancer J Clin 2005;55:74-108. Bruix J, Sherman M, Llovet JM, Beaugrand M, Lencioni R, Burroughs AK, et al. Clinical management of hepatocellular carcinoma. Conclusions of the Barcelona-2000 EASL conference. European Association for the Study of the Liver. J Hepatol 2001;35:421-430. Fattovich G, Stroffolini T, Zagni I, Donato F. Hepatocellular carcinoma in cirrhosis: incidence and risk factors. Gastroenterology 2004;127:S35- S50.